CLINICAL TRIAL: NCT03306667
Title: Clinical Pharmacology Study of FYU-981 for Subjects With Hepatic Insufficiency
Brief Title: Clinical Pharmacology of FYU-981 (Subjects With Hepatic Insufficiency)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Collaborators: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-015
Record Dates: First submitted 2017-09-20; First posted 2017-10-11 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Hepatic Insufficiency; Healthy
MeSH Terms: conditions — Hepatic Insufficiency | interventions — dotinurad

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal group (Experimental): Healthy control subjects
  Interventions: Drug: FYU-981
- Mild hepatic-insufficient group (Experimental): Patients with mild hepatic impaired function (Child-Pugh A)
  Interventions: Drug: FYU-981
- Moderate hepatic-insufficient group (Experimental): Patients with moderate hepatic impaired function (Child-Pugh B)
  Interventions: Drug: FYU-981
- Severe hepatic-insufficient group (Experimental): Patients with severe hepatic impaired function (Child-Pugh C)
  Interventions: Drug: FYU-981

INTERVENTIONS:
Drug: FYU-981 — Oral single dosing

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, pharmacodynamics and safety after single oral administration of FYU-981 to subjects with hepatic insufficiency and with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy subjects or adult cirrhosis patients
* Body mass index: >=18.5 and <30.0

Exclusion Criteria:

* Subjects with any disease or any history of diseases that might be unsuitable for participation in the clinical study (except for cirrhosis patients with hepatic diseases)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax: Maximum plasma concentration) | 48 hours
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 48 hours
Pharmacokinetics (T1/2: Elimination half-life of plasma concentration) | 48 hours
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 48 hours
Pharmacokinetics (CLtot/F: Total clearance / Fraction of dose absorbed) | 48 hours
Pharmacokinetics (kel: Elimination rate constant) | 48 hours
Pharmacokinetics (Vd/F: Distribution volume / Fraction of dose absorbed) | 48 hours
Pharmacokinetics (MRT: Mean residence time) | 48 hours
Pharmacodynamics (Serum concentration of uric acid) | 48 hours
Pharmacodynamics (Amount of uric acid excreted in urine) | 48 hours
Safety (Incidence of treatment-emergent adverse events) | 192 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Matsumoto, Study Director — Clinical Research Department
Locations (1):
- Mochida Investigational sites, Tokyo, Japan